CLINICAL TRIAL: NCT02561039
Title: Randomized, Open Label Study to Assess the Efficacy and Safety of the Intravenous and Oral Ibandronic Acid for Improving the Performance Status of Patients With Malignant Bone Disease Secondary to Solid Tumors and Hematological Malignancies
Brief Title: A Study of Ibandronate (Bondronat) in Participants With Malignant Bone Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20713
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pain; Bone Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid

ARMS (2):
- Ibandronate IV Infusion (Experimental): Participants will receive ibandronate, 6 mg via IV infusion, every 3 to 4 weeks for 4 months.
  Interventions: Drug: Ibandronate
- Ibandronate PO Tablet (Experimental): Participants will receive ibandronate, 50 mg PO daily, for 4 months.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Participants will receive ibandronate, either as a 6-mg IV infusion every 3 to 4 weeks or a 50-mg tablet PO daily, for 4 months.
  Other Names: Bondronat

SUMMARY:
This study will assess the efficacy and safety of ibandronate (Bondronat), administered intravenously (IV) or orally (PO), in participants with malignant bone disease and moderate to severe pain. Participants will be randomized to receive ibandronate either as a 6-mg IV infusion every 3 to 4 weeks or a 50-mg tablet PO daily. Pain response and Karnofsky Performance Index (KPI) will be measured at intervals throughout the study. The anticipated time on study treatment is 4 months and the target sample size is 150 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Malignant bone disease due to multiple myeloma or cancer of the lung, prostate, gastrointestinal (GI) tract, ovary, or bladder
* Bone pain defined as a Brief Pain Inventory (BPI) most acute pain score greater than or equal to 4
* Radiologically confirmed bone disease disease

Exclusion Criteria:

* Previous treatment with ibandronate (Bondronat) within previous 2 months
* Severely impaired renal function
* Known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Response rate according to reduction in BPI most acute pain score from Baseline | Month 4
Change in KPI | Baseline to Month 4

SECONDARY OUTCOMES:
Time to onset of decrease in most acute pain score | Up to 4 months
Analgesic consumption according to participant diary | Up to 5 months
Incidence of adverse events | Up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (7):
- Bulgaria (7):
  - Burgas
  - Haskovo
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Vratsa